CLINICAL TRIAL: NCT04703205
Title: A Placebo-controlled, Randomized, Double-blind Study in COvid-19 Patients With iveRmectin; An inVEstigator iniTiaTEd Trial
Brief Title: Study in COvid-19 Patients With iveRmectin (CORVETTE-01)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kitasato University (Other)
Responsible Party: Principal Investigator, KUNIHIRO YAMAOKA, KitasatoUniversity SchoolofMedicine Professor, Kitasato University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORVETTE-01
Record Dates: First submitted 2020-12-01; First posted 2021-01-11 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ivermectin (Experimental): Ivermectin group: Ivermectin approximately 200 μg/kg administered as a single oral dose on Day 1 (fasting state) subjects take the study drug (3 mg tablet of ivermectin) at the dose of the study drug taken once per body weight of the subject.
  Interventions: Drug: Ivermectin 3 MG
- placebo (Placebo Comparator): Placebo group: Placebo without ivermectin as an ingredient, single oral administration on Day 1 (fasting state) the control drug (ivermectin placebo tablet) at the dose of the study drug taken once per body weight of the subject.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin 3 MG — Ivermectin approximately 200 μg/kg administered as a single oral dose on Day 1 (fasting state)
  Arms: ivermectin
Drug: Placebo — Placebo group: Placebo without ivermectin as an ingredient, single oral administration on Day 1 (fasting state)
  Arms: placebo

SUMMARY:
Treatment of mild COVID-19 is basically performed at an outpatient clinic, then when the symptom and clinical findings exacerbate to a moderate level, patients are admitted. There is no standard treatment for mild cases. This study will investigate whether ivermectin administration suppresses the replication of SARS-CoV-2 in mild to moderate COVID-19 by investigating the negative rate of SARS-CoV-2 PCR by a randomized controlled trial. Subjects are assigned to two groups, the placebo group, and the ivermectin group. The target number of each treatment arm is 120, a total of 240 cases. A single oral administration of 200 ㎍/kg of ivermectin or an ivermectin-free placebo will be administered on an empty stomach. Time to negativization of SARS-CoV-2 PCR as the primary endpoint with additional efficacy and safety of the process will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. A person who has been diagnosed with COVID-19 (including asymptomatic) by the COVID-19 PCR test (SARS-CoV-2 nucleic acid detection) within 3 days before the qualification test.
2. A person with oxygen saturation (SpO2) in the room air of 95% or more.
3. A person who are 20 years or older at the time of obtaining consent.
4. A person who weigh 40 kg or more at the time of qualification test.
5. A person who understands the content of this clinical trial and can obtain written consent to participate in the clinical trial.

Exclusion Criteria:

1. A woman who is in lactation period or who may be pregnant, or those who do not agree to prevent pregnancy by medically appropriate means for up to 7 days after study drug administration.

   Medically appropriate contraception means that using a combination of two or more of the following: not having sexual intercourse, taking surgical sterilization such as vasectomy or intrauterine device, taking oral contraceptive, using condom.
2. A person who has severe liver damage (AST or ALT at the time of qualification test is more than 3 times the upper limit of institutional standard and total bilirubin is more than twice the upper limit of institutional standard value), renal disorder (eGFR of eligibility test value 30 mL/min/1.73m2 or less).
3. A person with hypersensitivity to ivermectin.
4. A person with a history of severe drug allergies such as Stevens-Johnson syndrome, toxic epidermal necrolysis.
5. A person who has received the prohibited medication within the past month (within the past 6 months for biologics), or those who need to use the prohibited medication during the clinical trial period.
6. Those who are scheduled to receive SARS-CoV-2 vaccination from the date of consent to the end of the follow-up period.
7. A person who are currently participating in other clinical trials or who have participated in other clinical trials within 30 days before obtaining consent.
8. In addition, a person who is determined to be unsuitable as a subject of this clinical trial by the principal investigator."

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 PCR test (SARS-CoV-2 nucleic acid detection) Period until the COVID-19 PCR test (SARS-CoV-2 nucleic acid detection) becomes negative | 15days
  Period until the COVID-19 PCR test (SARS-CoV-2 nucleic acid detection) becomes negative

CONTACTS AND LOCATIONS:
Overall Officials: Kunihiro K.Y Yamaoka, Ph.D, Principal Investigator — Kitasato University Hospital
Locations (1):
- Kitasato University, Sagamihara, Kanagawa, Japan

REFERENCES:
- [Background] Nicolas P, Maia MF, Bassat Q, Kobylinski KC, Monteiro W, Rabinovich NR, Menendez C, Bardaji A, Chaccour C. Safety of oral ivermectin during pregnancy: a systematic review and meta-analysis. Lancet Glob Health. 2020 Jan;8(1):e92-e100. doi: 10.1016/S2214-109X(19)30453-X. PMID 31839144
- [Background] Lv C, Liu W, Wang B, Dang R, Qiu L, Ren J, Yan C, Yang Z, Wang X. Ivermectin inhibits DNA polymerase UL42 of pseudorabies virus entrance into the nucleus and proliferation of the virus in vitro and vivo. Antiviral Res. 2018 Nov;159:55-62. doi: 10.1016/j.antiviral.2018.09.010. Epub 2018 Sep 26. PMID 30266338
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Rajter JC, Sherman MS, Fatteh N, Vogel F, Sacks J, Rajter JJ. Use of Ivermectin Is Associated With Lower Mortality in Hospitalized Patients With Coronavirus Disease 2019: The Ivermectin in COVID Nineteen Study. Chest. 2021 Jan;159(1):85-92. doi: 10.1016/j.chest.2020.10.009. Epub 2020 Oct 13. PMID 33065103
- [Derived] Wada T, Hibino M, Aono H, Kyoda S, Iwadate Y, Shishido E, Ikeda K, Kinoshita N, Matsuda Y, Otani S, Kameda R, Matoba K, Nonaka M, Maeda M, Kumagai Y, Ako J, Shichiri M, Naoki K, Katagiri M, Takaso M, Iwamura M, Katayama K, Miyatsuka T, Orihashi Y, Yamaoka K; CORVETTE-01 Study Group. Efficacy and safety of single-dose ivermectin in mild-to-moderate COVID-19: the double-blind, randomized, placebo-controlled CORVETTE-01 trial. Front Med (Lausanne). 2023 May 22;10:1139046. doi: 10.3389/fmed.2023.1139046. eCollection 2023. PMID 37283627